CLINICAL TRIAL: NCT01984450
Title: A Study to Compare Two Articular Cartilage Repair Techniques in the Knee Joint: Autologous Collagen Induced Chondrogenesis (ACIC) Vs. Mesenchymal Cell Induced Chondrogenesis (MCIC).
Brief Title: A Study to Compare Two Techniques for Articular Cartilage Repair:ACIC Vs. MCIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shetty-Kim Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKRF 002
Record Dates: First submitted 2013-10-11; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Articular Cartilage Defect
Keywords: Articular cartilage; Autologous collagen; BMAC
MeSH Terms: interventions — Acyclovir; Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACIC (Active Comparator): The patients in this group will be treated by the ACIC technique, which uses autologous collagen to regenerate articular cartilage. ACIC is a single stage arthroscopic procedure. It is done as a day case procedure. The cartilage defect is debrided and implanted with a collagen + fibrin gel mixture under CO2 insufflation.
  Interventions: Procedure: ACIC; Device: implant with a collagen + fibrin gel mixture
- MCIC (Active Comparator): The patients in this group will be treated by the MCIC technique, which uses concentrated BMAC to regenerate articular cartilage. MCIC is a single stage arthroscopic procedure. It is done as a day case procedure. BMAC is harvested intraoperatively and concentrated. It is then mixed with a fibrin gel and implanted under CO2 insufflation.
  Interventions: Procedure: MCIC

INTERVENTIONS:
Procedure: ACIC — Autologous Collagen Induced Chondrogenesis (ACIC):
  ACIC is a single stage arthroscopic procedure. It is done as a day case procedure. The cartilage defect is debrided and implanted with a collagen + fibrin gel mixture under CO2 insufflation.
  Arms: ACIC
Procedure: MCIC — Mesenchymal Cell Induced Chondrogenesis (MCIC):
  MCIC is a single stage arthroscopic procedure. It is done as a day case procedure. BMAC is harvested intraoperatively and concentrated. It is then mixed with a fibrin gel and implanted under CO2 insufflation.
  Arms: MCIC
Device: implant with a collagen + fibrin gel mixture
  Arms: ACIC

SUMMARY:
Study Title: A study to compare two articular cartilage repair techniques in the knee joint: Autologous Collagen Induced Chondrogenesis (ACIC) Vs. Mesenchymal Cell Induced Chondrogenesis (MCIC).

Study hypothesis: We start with the hypothesis that both treatments are equally effective.

Trial Design: This is a prospective study. The participating patients will be divided into two groups, each group receiving either one of the treatment modalities. This study will not be randomised or blinded. Both procedures will be done at the Spire Alexandra Hospital by Professor A. A Shetty, who is one half of the team that devised both techniques.

Trial Participants: All participants will be from patients attending Professor Shetty's clinic at the Spire Alexandra Hospital.

Planned Sample Size: 50 patients in each arm.

Follow-up duration: The participating patients will be followed up at 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years following the surgery by visits to the clinic and assessed clinically. The surgical outcomes will be measured by by IKDC, KOOS and Lysholm scores; cartilage growth will be measured by the MOCART score.

Planned Trial Period: Two to three years

Primary Objective: To establish superiority, if any, of either procedure over the other.

Primary Endpoint: At the end of the 2 year follow up for all participating patients.

DETAILED DESCRIPTION:
BACKGROUND: Articular cartilage repair in the knee is aimed at young patients with area(s) of cartilage loss and no deformity of the knee. These patients aren't indicated for a knee replacement. Articular cartilage repair leads to improvement of symptoms of pain, locking and function. Traditionally, articular cartilage repair has always involved exposing the entire knee joint with an arthrotomy. This, though effective, would lead to a large scar, longer hospital stay, longer rehabilitation and its associated complications. Also, the use of Bone Marrow Aspirate Cells (BMAC) for the purpose of cartilage repair has long been debated with both sides having valid arguments and good surgical results.

RATIONALE: Both procedures in this study are performed in one stage, arthroscopically and as day case procedures, which offers minimal scarring and quicker recovery. This automatically confers a significant advantage over the traditional surgical techniques.

To correct the articular cartilage defect, the ACIC method requires autologous Atellocollagen (a protein based structure), while the MCIC method uses concentrated BMAC taken from the patient's iliac crest.

Both procedures have shown encouraging results in terms of pain relief, cartilage growth and improved function. Since one technique utilises a protein based reagent and the other involves mesenchymal cells, this study aims to ascertain if either technique is superior to the other.

STUDY DESIGN: This study aims to compare two techniques of articular cartilage repair in the knee, namely Autologous Collagen Induced Chondrogenesis (ACIC) and Mesenchymal Cell Induced Chondrogenesis (MCIC). The principal objective of is to ascertain and assess the superiority, if any, of either surgical technique over the other. The superiority will be assessed with by the certain scoring systems (IKDC, KOOS, Lysholm and MOCART) measured pre- and post-operatively.

Depending on which procedure the patient chooses to have, they will be allotted to either the ACIC or the MCIC group. The patient is followed up in the clinic at the Spire Alexandra Hospital at 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years following the surgery and their progress is documented by questionnaires and clinical examination. MRI scans are done at one and two years to assess the extent of cartilage growth.

SURGICAL TECHNIQUES

Autologous Collagen Induced Chondrogenesis (ACIC):

ACIC is a single stage arthroscopic procedure. It is done as a day case? procedure and the patient is admitted a few hours before the procedure. The anaesthetic method depends is the Anaesthesiologist's prerogative and depends on the patient's general health. Under sterile conditions in an operating theatre, the arthroscopic instruments are introduced inside the knee joint. As assessed previously by MRI scans, the area of cartilage defect is debrided by curettage, shaving and burring and then microfractured. The ACIC method utilises autologous Atellocollagen, a protein based structure, mixed with thrombin and fibrinogen to form a gel which coats the area with a cartilage defect. The entry ports are then closed and the knee is covered with a sterile dressing. The patient is transferred to the surgical recovery ward and, when medically stable, then transferred to their room on the ward.

After discharge from the hospital, the patient is advised partial weight bearing on the operated leg for 6 weeks after the surgery. They also undergo 5 sessions of physiotherapy. Surgical clips and sutures are removed at 2 weeks following the surgery.

Mesenchymal Cell Induced Chondrogenesis (MCIC):

MCIC is a single stage arthroscopic procedure. It is done as a day case? procedure and the patient is admitted a few hours before the procedure. The anaesthetic method depends is the Anaesthesiologist's prerogative and depends on the patient's general health. Under sterile conditions in an operating theatre, the arthroscopic instruments are introduced inside the knee joint. As assessed previously by MRI scans, the area of cartilage defect is debrided by curettage, shaving and burring and then microfractured. The MCIC method involves aspiration of Bone Marrow Aspirate Cells (BMAC) from the patient's iliac crest (hip bone) and concentrating the cells by centrifugation in the operation theatre itself. The BMAC are then mixed with thrombin and fibrinogen to form a gel which coats the area with a cartilage defect.

After discharge from the hospital, the patient is advised partial weight bearing on the operated leg for 6 weeks after the surgery. They also undergo 5 sessions of physiotherapy. Surgical clips and sutures are removed at 2 weeks following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years to 65 years.
* Diagnosed with articular cartilage defect in the knee (ICRS/Outerbridge grade III/IV cartilage lesions as assessed on MRI scan).
* No other significant medical co-morbidities, as assessed by pre-operatively, that could interfere with surgery results of trial eg. Hypertension, COPD etc.
* Participant has clinically acceptable laboratory and ECG tests at pre-assessment clinic.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Up to 3 lesions of sizes 2-8 square cm.

Exclusion Criteria:

* Generalized and/or inflammatory arthritis
* Active joint inflammation
* More than 5 degrees of varus or valgus deformity
* Age below 18 and over 65 years
* More than 4 lesions
* Lesions more than 8 square cm.
* Significant co-morbidities or classified as ASA grade 3/4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 2 years
  This study aims to compare two techniques of articular cartilage repair in the knee, namely Autologous Collagen Induced Chondrogenesis (ACIC) and Mesenchymal Cell Induced Chondrogenesis (MCIC). The principal objective of is to ascertain and assess the superiority, if any, of either surgical technique over the other. The superiority will be assessed with by the IKDC score measured pre- and post-operatively
Radiological outcome | 2 years
  This study aims to compare two techniques of articular cartilage repair in the knee, namely Autologous Collagen Induced Chondrogenesis (ACIC) and Mesenchymal Cell Induced Chondrogenesis (MCIC). The principal objective of is to ascertain and assess the superiority, if any, of either surgical technique over the other. The superiority will be assessed with by the MOCART score measured pre- and post-operatively
Clinical outcome | 2 years
  This study aims to compare two techniques of articular cartilage repair in the knee, namely Autologous Collagen Induced Chondrogenesis (ACIC) and Mesenchymal Cell Induced Chondrogenesis (MCIC). The principal objective of is to ascertain and assess the superiority, if any, of either surgical technique over the other. The superiority will be assessed with by the KOOS score measured pre- and post-operatively
Clinical outcome | 2 years
  This study aims to compare two techniques of articular cartilage repair in the knee, namely Autologous Collagen Induced Chondrogenesis (ACIC) and Mesenchymal Cell Induced Chondrogenesis (MCIC). The principal objective of is to ascertain and assess the superiority, if any, of either surgical technique over the other. The superiority will be assessed with by the Lysholm score measured pre- and post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Asode A Shetty, MD, PhD, MCh, FRCS, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Kent Knee Unit, Walderslade, Kent, United Kingdom